CLINICAL TRIAL: NCT00927056
Title: Early Activity Monitoring and Pain Assessment in Minimally Invasive Microdiscectomy Versus Conventional Open Microdiscectomy For The Treatment of Lumbar Herniated Disc
Brief Title: Evaluation of Minimally Invasive Microdiscectomy Versus Conventional Open Microdiscectomy For Lumbar Herniated Disc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Michael Johnson/Principal Investigator, Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2006:186
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Lumbar Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Minimally Invasive Microdiscectomy (Active Comparator)
  Interventions: Procedure: Microdiscectomy
- Conventional Open Microdiscectomy (Active Comparator)
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: Microdiscectomy — Minimally invasive microdiscectomy versus conventional open microdiscectomy

SUMMARY:
Overall Objective: To evaluate pain and functional status of patients undergoing surgical correction for lumbar herniated disc, pre- and post-surgery, using subjective (VAS, Oswestry, PSQI, Patient Expectation), as well as, objective measures of physical activity (triaxial accelerometry).

Design and Methods: Two groups of subjects will be examined; 1) patients diagnosed with lumbar herniated disc undergoing minimally invasive microdiscectomy (MD), and 2) patients diagnosed with lumbar herniated disc undergoing open microlumbar discectomy (OD).

Subjects who agree to participate, will be assessed (assessments listed below) after the diagnosis and prior to surgery. The subject will then be assessed postop and they will continue with follow-up after surgery with a visit at 3 weeks postop. Both methods of discectomy will be discussed with the subject. Once the subject has consented to participate (and prior to surgery), subjects will be randomized with a 50/50 chance of being placed in the MD or OD groups. Subjects will be distributed into the MD group and the OD group using a block randomization method. The study will be single blinded. A longitudinal, within group, comparison will be made to assess the change in the measured parameters. Data involving the MD and OD groups will be accumulated in a cross-sectional fashion.

Subjects will be recruited from the referrals to the practices of the Orthopedic and Neurosurgeon Spine Surgeons at the Health Sciences Centre. This encompasses the majority of new and currently managed cases in the Manitoba and Northwestern Ontario.

Subjects will be between the ages of 18 and 90. Male and female subjects will be recruited into the study. All patients will clinically demonstrate unilateral lower extremity pain in greater proportion to low back pain symptoms if present. Imaging (CT) will document single level lumbar herniated nucleus pulposis. Exclusion criteria will be cauda equina syndrome, progressive neurologic deficit, bilateral lower extremity symptoms, low back pain more than leg pain, the existence of significant co-morbidity (e.g. cardiac condition, disease, etc.) of any form, and any other physical limitations (musculoskeletal injury). Subjects participating will be required to speak and read English.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 18 and 90.
* Male and female subjects will be recruited into the study.
* All patients will clinically demonstrate unilateral lower extremity pain in greater proportion to low back pain symptoms if present. Imaging (CT) will document single level lumbar herniated nucleus pulposis.
* Subjects participating will be required to speak and read English.

Exclusion Criteria:

* Cauda equina syndrome, progressive neurologic deficit, bilateral lower extremity symptoms, low back pain more than leg pain, the existence of significant co-morbidity (e.g. cardiac condition, disease, etc.) of any form, and any other physical limitations (musculoskeletal injury).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Physical activity monitor | continuous for 3 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Johnson, MD, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Spine Research Lab, Winnipeg, Manitoba, Canada